CLINICAL TRIAL: NCT03318874
Title: Comparing the Effects of THERA°PEARL Eye Mask (Bausch & Lomb Inc., New York, USA) With the Use of Blephasteam® (Spectrum Thea Pharmaceuticals LTD, Macclesfield, UK).
Brief Title: Optimization of the Treatment of Dry Eye Disease Caused by Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Schepens Eye Research Institute (Other); The Norwegian Dry Eye Clinic (Other Government)
Responsible Party: Principal Investigator, Jonatan Olafsson, Medical Student, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/1983
Record Dates: First submitted 2017-10-04; First posted 2017-10-24 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction
Keywords: Dry Eye Disease; Meibomian Gland Dysfunction; Blephasteam; THERA°PEARL Eye Mask
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blephasteam (Experimental): Heat delivery device, to be used according to guidelines from manufacturer.
  Interventions: Device: Blephasteam; Drug: Hylo-comod
- THERA°PEARL Eye Mask (Active Comparator): Heat delivery device, to be used according to guidelines from manufacturer.
  Interventions: Device: THERA°PEARL Eye Mask; Drug: Hylo-comod

INTERVENTIONS:
Device: Blephasteam — Steam delivery goggles, once daily
  Arms: Blephasteam
Device: THERA°PEARL Eye Mask — Heat delivery device, delivering heat to the eyelids, once daily
  Arms: THERA°PEARL Eye Mask
Drug: Hylo-comod — Tear substitute containing hyaluronic acid, four times daily
  Other Names: Sodium hyaluronate

SUMMARY:
An open label, randomized controlled study in a Norwegian population with meibomian gland dysfunction. Patients will be randomized to one of two groups: THERA°PEARL Eye Mask (Bausch & Lomb Inc., New York, USA) or Blephasteam® (Spectrum Thea Pharmaceuticals LTD, Macclesfield, UK). All patients will receive Hylo-comod (URSAPHARM Arzneimittel GmbH, Saarbrücken, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Meibomian Gland Dysfunction
* Eligible for heat treatment
* Ocular Surface Disease Index (OSDI) >12
* Quality or expressibility score ≤20 years old: >1 or >20 years old: ≥1
* Non-invasive tear film break-up time (NITBUT) <10 s in at least one eye
* Schirmer-1 test >5 mm after 5 min

Exclusion Criteria:

* Glaucoma,
* Ocular allergy
* Autoimmune disease
* Contact lens-wear during study
* Current punctal plugging
* Pregnant/lactating
* Candidate for topical anti-inflammatory
* Cicatricial meibomian gland dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Tear film break-up time | Change from baseline at three and six months
  Fluorescein applied to tear film, time measured until tear film breaks up after blink. Range of scale from 1 second and higher, where higher values are considered preferable for the patients. Values under 10 seconds are indicative for dry eye disease.

SECONDARY OUTCOMES:
Ocular Surface Disease Index | Change from baseline at three and six months
  Dry Eye Self reported Questionnaire, score ranging from 0-100, where lower values are considered preferable for the patients, indicating less symptoms. Values over 12 are indicative for dry eye disease.
McMonnies Questionnaire | Change from baseline at three and six months
  Dry Eye Self reported Questionnaire. Index ranges from 0 to 45, where a higher score is regarded as more indicative of dry eye disease. A cut-point of greater than 14.5 is recommended for a dry eye diagnosis.
Ocular surface staining Ocular surface staining | Change from baseline at three and six months
  Fluorescein applied to tear film, staining scored after the Oxford staining scheme, values ranging from 0-15, lower values are considered better for the patient.
Tear cytokine levels | Change from baseline at three and six months
  Multiplex analysis of tear fluid
Schirmer's test | Change from baseline at three and six months
  Measurement of 5 minutes of tear production, values ranging from 0 and higher, where lower values are considered worse for the patient. Values under 5 mm are indicative for dry eye disease.
Meibum Quality | Change from baseline at three and six months
  Guidelines based on MGD-report of 2011, values ranging from 0-24, where lower values are considered better for the patient, indicating the quality of the meibum secretion.
Meibum Expressibility | Change from baseline at three and six months
  Guidelines based on MGD-report of 2011, values ranging from 0-3, where lower values are considered better for the patient, indicating open meibomian glands.
Tear osmolarity | Change from baseline at three and six months
  Osmolarity measured with TearLab, where values under 300 mOsml/L are considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Tor P Uthiem, MD, Phd., Principal Investigator — Oslo University Hospital
Locations (1):
- The Norwegian Dry Eye Clinic, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Olafsson J, Lai X, Landsend ECS, Olafsson S, Parissi E, Utheim OA, Raeder S, Badian RA, Lagali N, Dartt DA, Utheim TP. TheraPearl Eye Mask and Blephasteam for the treatment of meibomian gland dysfunction: a randomized, comparative clinical trial. Sci Rep. 2021 Nov 17;11(1):22386. doi: 10.1038/s41598-021-01899-8. PMID 34789807

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT03318874/Prot_SAP_000.pdf